CLINICAL TRIAL: NCT01509261
Title: A Phase Ⅲ Multi-center, Randomized, Double-blind, Active-controlled Study to Evaluate the Efficacy and Safety of Ilaprazole (20mg QD) in Adult Patients With Erosive Esophagitis
Brief Title: Efficacy Study of Ilaprazole to Treat Erosive Esophgitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IY-81149-EE03
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Erosive Esophagitis; GERD
Keywords: Erosive Esophagitis; Ilaprazole; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ilaprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ilaprazole (Experimental): Ilaprazole 20mg
  Interventions: Drug: Ilaprazole
- lansoprazole (Active Comparator): lansoprazole 30mg
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Ilaprazole — 20mg/Tap, QD
  Other Names: Noltec
  Arms: Ilaprazole
Drug: Lansoprazole — 30mg/Tap, QD
  Arms: lansoprazole

SUMMARY:
This study compared Ilaprazole 20mg with lansoprazole 30mg for the healing of erosive esophagitis and resolution of heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed erosive esophagitis as defined by the Los Angeles (LA) Classification Grading System (A-D) within 14 days prior to baseline.
* Episodes of heartburn or regurgitation has experienced during the last 7 days prior to baseline.

Exclusion Criteria:

* Coexisting diseases affecting the esophagus (eg, eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus. Presence of a Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) or Barrett's esophagus were not exclusionary.
* Current or a history of Zollinger-Ellison syndrome and other acid hypersecretory conditions, or current gastric or duodenal ulcer.
* Known hypersensitivity to any PPI (including lansoprazole, omeprazole, rabeprazole, pantoprazole or esomeprazole), any component of ilaprazole, or Gelusil.
* Cancer (except basal cell carcinoma of the skin) within 5 years prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The crude healing rate of EE at Week 8 of treatment as assessed by endoscopy | 8 Weeks
  Endoscopic healing of erosive esophagitis is defined as those participants who have endoscopically confirmed EE of Grade O as defined by the Los Angeles (LA) Classification Grading System. The definitions of each grade are: Grade O (No mucosal break), Grade A (Mucosal break <5 mm), Grade B (Mucosal break ≥5 mm), Grade C (Mucosal break continuous between two or more folds and <75% of the circumference) and Grade D (Mucosal break ≥75% of the circumference).

SECONDARY OUTCOMES:
The crude healing rate of EE at Week 8 of treatment as assessed by endoscopy | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim JinHo, Principal Investigator — Asan Medical Center
Locations (1):
- Local Institution, Seoul, South Korea